CLINICAL TRIAL: NCT03937765
Title: The Effect of Platelet Rich Plasma on Pain at Skin Graft Donor Sites
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Suspended per IRB
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRP Study
Record Dates: First submitted 2019-04-29; First posted 2019-05-06 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Skin Graft (Allograft) Rejection; Skin Graft Complications; Skin Graft Detachment; PRP
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Intervention Model Description: Each patient that will be undergoing a skin graft surgery will be randomized into either the PRP (intervention) group or the control group. Follow up and dressing changes will be the same for both groups. Each group will be prescribed a multi-modal pain regimen to reduce narcotic usage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP (Experimental): Intervention group will receive PRP instead of the standard of care for skin grafts. PRP Group-will remove surgical dressing post operative day 5. Donor site will be cleaned with soap and water daily and dressed with gauze daily until drainage stops.
  Interventions: Procedure: PRP harvest and preparation
- Control (No Intervention): Control group receiving the standard of care for skin grafts. Control Group-will remove gauze dressing post operative day 2 but leave adeptic. Donor site will be cleaned daily with soap and water. Gauze applied daily as needed for drainage and will be stopped when drainage stops. The adeptic, which forms a biologic dressing, will be removed by the patient over time as it lifts from the wound.

INTERVENTIONS:
Procedure: PRP harvest and preparation — The PRP harvest and preparation will be done in the operating room with the help of the hospital blood bank. The skin graft surgery will be completed by Dr. Jason Lowe and/or one of the Orthopaedic Surgery residents. Follow up will also be completed by Dr. Lowe or one of the residents. Data analysis will be done by Drs. Lowe and Manoharan.
  Each patient that will be undergoing a skin graft surgery will be randomized into either the PRP (intervention) group or the control group. Follow up and dressing changes will be the same for both groups. Each group will be prescribed a multi-modal pain regimen to reduce narcotic usage.
  Arms: PRP

SUMMARY:
The purpose of this study is to compare post-operative skin graft donor site pain between those treated with standard wound care vs PRP. Secondarily the study is designed to compare time to complete donor site healing. The null hypothesis is that here is no difference in post-operative donor site pain between those treated with standard wound care and PRP. The secondary null hypothesis is that there is no difference in time to donor site healing.

DETAILED DESCRIPTION:
A well-known complaint after a split thickness skin graft surgery is pain at the graft donor site. In our patients, it has been have noticed those whose donor sites have been treated with platelet rich plasma (PRP) have endorsed decreased pain compared to those who have not. During our literature review few studies have looked at this issue. One such study by Miller et. al. looked at 5 patients whose donor site was treated with PRP showed a significant decrease in pain on a Likert visual pain scale. Kakudo et al. performed a side-by-side comparison on a single patient with half the wound treated with PRP and the other as a control. They found better epithelization and reduced pain during dressing changes for the treatment group. Both of these studies show promising results for pain reduction with PRP use, unfortunately there are no high quality randomized control trials that have looked at this. Another issue is many studies on PRP assess reduction of pain as a secondary outcome and instead focus on wound healing and epithelization primarily.

This study hopes to elucidate the effect of PRP application on graft donor site pain. Patients will be recruited to the study and randomized into either treatment or control group based on medical necessity for a skin graft. This study will assess pain at the donor site via Likert pain scale and monitor narcotic pain medication use.

ELIGIBILITY:
Inclusion Criteria:

* Any patient requiring a split thickness skin graft and is above the age of 18.

Exclusion Criteria:

* Medical history of chronic pain at the donor site
* Inability to follow up
* Unable to participate in pre or post operative questionnaire inclusive of organic
* Traumatic, chemical or degenerative causes of altered mental sensorium
* Age <18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Patient post-operative donor site pain. | Through study completion, an average of 1 year
  Donor site pain according to the visual analog scale score. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."
Duration of donor site wound | Through study completion, an average of 1 year
  Duration of wound care after surgery
Opioid consumption | Through study completion, an average of 1 year
  Opioid consumption after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Aditya Manoharan, MD, Principal Investigator — University of Arizona College of Medicine Department of Orthopaedic Surgery; Jason Lowe, MD, Principal Investigator — University of Arizona College of Medicine Department of Orthopaedic Surgery
Locations (1):
- University of Arizona College of Medicine, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Miller JD, Rankin TM, Hua NT, Ontiveros T, Giovinco NA, Mills JL, Armstrong DG. Reduction of pain via platelet-rich plasma in split-thickness skin graft donor sites: a series of matched pairs. Diabet Foot Ankle. 2015 Jan 22;6:24972. doi: 10.3402/dfa.v6.24972. eCollection 2015. PMID 25623477
- [Result] Kakudo N, Kushida S, Minakata T, Suzuki K, Kusumoto K. Platelet-rich plasma promotes epithelialization and angiogenesis in a splitthickness skin graft donor site. Med Mol Morphol. 2011 Dec;44(4):233-6. doi: 10.1007/s00795-010-0532-1. Epub 2011 Dec 17. PMID 22179187
- [Result] Carter MJ, Fylling CP, Parnell LK. Use of platelet rich plasma gel on wound healing: a systematic review and meta-analysis. Eplasty. 2011;11:e38. Epub 2011 Sep 15. PMID 22028946
- [Result] Boonstra AM, Schiphorst Preuper HR, Reneman MF, Posthumus JB, Stewart RE. Reliability and validity of the visual analogue scale for disability in patients with chronic musculoskeletal pain. Int J Rehabil Res. 2008 Jun;31(2):165-9. doi: 10.1097/MRR.0b013e3282fc0f93. PMID 18467932
- [Result] Delgado DA, Lambert BS, Boutris N, McCulloch PC, Robbins AB, Moreno MR, Harris JD. Validation of Digital Visual Analog Scale Pain Scoring With a Traditional Paper-based Visual Analog Scale in Adults. J Am Acad Orthop Surg Glob Res Rev. 2018 Mar 23;2(3):e088. doi: 10.5435/JAAOSGlobal-D-17-00088. eCollection 2018 Mar. PMID 30211382